CLINICAL TRIAL: NCT01156285
Title: Acute Anterior Uveitis: Psychic Burden and Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Hietzing (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Saskia M Maca, MD, Hospital Hietzing
Other Study IDs: MAC110
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Anterior Uveitis
MeSH Terms: conditions — Uveitis, Anterior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AAU: patient with acute attack of anterior uveitis
  Interventions: Other: Filling in a patient questionnaire

INTERVENTIONS:
Other: Filling in a patient questionnaire — Filling in a patient questionnaire

SUMMARY:
Acute anterior uveitis (AU) is a common reason for attendance at ophthalmic outpatient clinics. The painfulness and the fear of a transient or even persistent loss of vision may markedly reduce the individual's subjective well-being and pose a psychological burden.

This study will test the hypothesis that during an attack of AU the patient experiences a marked reduction in psychological and physical well-being.

Prospective, hospital-based epidemiologic study using a patient questionnaire with standardized psychological tests and a pain scale.

ELIGIBILITY:
Inclusion Criteria:

* Acute attack of anterior uveitis

Exclusion Criteria:

* Other forms of uveitis
* Chronic anterior uveitis
* Therapy started

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute attack of anterior uveitis
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2010-05; Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Saskia M Maca, MD, Study Director — Hospital Hietzing
Locations (2):
- Austria (2):
  - Department of Ophthalmology, Medical University Graz, Graz, Styria
  - Department of Ophthalmology, Hietzing Hospital, Vienna, Vienna